CLINICAL TRIAL: NCT04285294
Title: Molecular Signatures of Cutaneous Squamous Cell Carcinoma During Recessive Dystrophic Epidermolysis Bullosa
Acronym: SIMOCEB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190820
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RDEB patients with a cSCC
- Non-RDEB patients with a SCC induced by ultraviolet radiation
- Healthy donors without RDEB nor SCC

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is a hereditary skin disease characterized by cutaneous and mucosa fragility. Blister formations and erosions, resulting in chronic wounds and dystrophic scars, lead development of aggressive cutaneous squamous cell carcinoma (cSCC) in young subjects. cSCC in RDEB patients are often recurrent and sometimes aggressive. Although fibrotic and inflammatory microenvironment plays an important role in the tumoral process, specific mechanisms in cSCC of RDEB patients are still unknown. Actually, the only treatment is a wide surgical excision with poor prognostic (80% of death after the first occurrence of cSCC).

The objective of the study is to describe the molecular signatures in the cSCC in RDEB patients

ELIGIBILITY:
Inclusion Criteria:

* for RDEB patients with a SCC :

  1. aged older than 18 years old
  2. one or more SCC surgically treated
  3. signed genetic consent form
* for non-RDEB patients with a SCC induced by ultraviolet radiation :

  1. aged older than 18 years old
  2. one or more SCC induced by ultraviolet radiation
  3. signed genetic consent form

Exclusion Criteria:

* under protection by law (tutorship or curatorship)
* without health insurance coverage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RDEB patients with a SCC and non-RDEB patients with a SCC induced by ultraviolet radiation
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Characterize the molecular signatures in the cSCC and the peri-tumoral dystrophic area occurring in RDEB patients | at inclusion
  Molecular signatures will be assessed by genomic, transcriptomic, and proteomic analyses

SECONDARY OUTCOMES:
Comparison of molecular signature according to the aggressive evolution | at inclusion
  Molecular signatures will be assessed by genomic, transcriptomic, proteomic analyses and will be compared between RDEB patients with different clinical outcomes (cSCC with an aggressive and metastatic evolution versus cSCC without aggressive evolution at 3 months).
Comparison of molecular signatures between cSCC from RDEB patients versus cSCC from non-RDEB patients (induced by ultraviolet radiation) | at inclusion
  Molecular signatures will be assessed by genomic, transcriptomic, and proteomic analyses and will be compared between cSCC from RDEB patients versus cSCC from non-RDEB patients (induced by ultraviolet radiation)